CLINICAL TRIAL: NCT06923384
Title: Screening and Brief Intervention for Prescription Stimulant Misuse and Diversion: Refining and Piloting a Curriculum for College Health Providers
Brief Title: SBI for PSM and PSD
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: California State University, Long Beach (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R34DA056596 (NIH); 1R34DA056596-01A1 (NIH)
Record Dates: First submitted 2025-04-04; First posted 2025-04-11 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Prescription Stimulant Misuse; Prescription Stimulant Diversion
Keywords: prescription stimulants

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three conditions: control, face-to-face intervention with trained providers, or e-Intervention that involves watching a video from a health provider and responding to questions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Placebo Comparator): Students complete the assessments at each time point, but do not receive any intervention or informational material.
  Interventions: Behavioral: Control
- F2F (Experimental): After T1 assessment, students meet with a trained provider and receive prevention or brief intervention. Students then complete assessments at two additional times.
  Interventions: Behavioral: F2F
- eSBI (Experimental): After T1 assessment, students watch and respond to a prevention or brief intervention video series. Students then complete assessments at two additional times.
  Interventions: Behavioral: eSBI

INTERVENTIONS:
Behavioral: F2F — After T1 assessment, students meet with a trained provider and receive prevention or brief intervention. Students then complete assessments at two additional times.
  Arms: F2F
Behavioral: eSBI — After T1 assessment, students watch and respond to a prevention or brief intervention video series. Students then complete assessments at two additional times.
  Arms: eSBI
Behavioral: Control — Students complete the assessments at each time point, but do not receive any intervention or informational material.
  Arms: Control

SUMMARY:
A pilot randomized controlled trial to assess the feasibility, acceptability, and impact of screening and brief intervention to address prescription stimulant misuse and diversion among college students.

DETAILED DESCRIPTION:
A screening and brief intervention including a control group, face-to-face group, and e-intervention group where the focus is prevention or brief intervention or referral to treatment related to students prescription stimulant misuse and diversion behaviors. Students will complete assessments at three time points, and the health providers who implement the intervention will also complete assessments.

ELIGIBILITY:
Inclusion Criteria:

Age 18 and student at the campus serving as the intervention site; Passive recruitment: Student has a scheduled appointment for a physical/wellness exam. Active recruitment: Student has a past 3 month history of PSM or PSD.

Exclusion Criteria:

Any eligible student who, during the course of the session, demonstrates the need for immediate mental health services, will have the study session terminated so that participant can receive needed care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-08-11 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Prescription Stimulant Misuse | 30 days
  Students report on their experience with prescription stimulant misuse behaviors. PSM is assessed at T1, pre-intervention, and T3, 30-Days post intervention.
Prescription Stimulant Diversion | 30 days
  Students report on their experience with prescription stimulant diversion behaviors. PSD is assessed at T1, pre-intervention, and T3, 30-Days post intervention.

SECONDARY OUTCOMES:
PSM Intentions | 30 days
  Intention to engage in PSM is measured at T1 (pre-intervention), T2 (immediate post), and T3 (30 Day post intervention)
PSD Intentions | 30 days
  Intention to engage in PSM is measured at T1 (pre-intervention), T2 (immediate post), and T3 (30 Day post intervention).

CONTACTS AND LOCATIONS:
Locations (1):
- CSULB, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual data will not be shared due to confidentiality agreements with participants, but study protocol, analysis plan, informed consent, and clinical study reports will be shared.